CLINICAL TRIAL: NCT01638416
Title: A Multi-centre Randomised Double Blinded Phase III Trial of the Effect of Standard Issue Red Blood Cell Blood Units on Mortality Compared to Freshest Available Red Blood Cell Units
Brief Title: Standard Issue Transfusion Versus Fresher Red Blood Cell Use in Intensive Care- A Randomised Controlled Trial
Acronym: TRANSFUSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Australian and New Zealand Intensive Care Research Centre (Other)
Collaborators: Australian Red Cross (Other); New Zealand Blood Service (Other); Irish Blood Transfusion Service (Other); Finnish Red Cross Blood Service (Other); King Abdulaziz Medical City (Other Government); University College Dublin (Other)
Responsible Party: Principal Investigator, David James Cooper, Professor, Australian and New Zealand Intensive Care Research Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANZICRCDJC006
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Transfusion; Age of Blood
MeSH Terms: interventions — Blood Transfusion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two staff not involved in the direct care of each patient checked the red-cell units, and concealed the collection and expiry dates from clinical staff using a bag with opaque panels (Australia, Ireland and Saudi Arabia), or an obscuring sticker (NZ and Finland).
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of care (Active Comparator): Blood Transfusion Standard of care- oldest blood.
  Interventions: Other: Blood transfusion
- Arm B (Other): Blood Transfusion Freshest blood.
  Interventions: Other: Blood transfusion

INTERVENTIONS:
Other: Blood transfusion — Blood transfusion in ICU patients aged 18 and over.

SUMMARY:
In Australia, blood for transfusion has a "use by" date of 42 days after collection. The actual age of blood given to patients depends on what is available at the time and the rate of usage. During the last decade, it has been reported that blood transfusion in patients admitted to intensive care was associated with an independent increase of mortality. Some research suggests that transfusion of fresher blood might help patients in the intensive care unit to reach a better recovery. This project will test whether patients who receive 'fresher' blood do better than patients who receive 'standard issue' blood.

DETAILED DESCRIPTION:
Inclusion criteria

•Patients hospitalised in ICU with an anticipated ICU stay of at least 24 hours, in whom the decision has been made by medical staff to transfuse at least one RBC unit.

Exclusion criteria

* Age younger than 18
* Previous RBC transfusion during the current hospital admission (including transfusion in another hospital for transferred patients)
* Diagnosis of transplantation or hematologic diseases
* Pregnancy
* Cardiac surgery during the present hospital admission
* Expected to die imminently (<24hrs)
* The treating physician believes it is not in the best interest of the patient to be randomised in this trial.
* Known objection to the administration of human blood products
* Participation in a competing study

Primary outcome- 90 day mortality

Secondary outcomes

1. 28 day mortality
2. Persistent Organ Dysfunction combined with death at 28
3. Days alive and free of mechanical ventilation at day 90 post randomisation
4. Day alive and free of renal replacement therapy at day 90 post randomisation
5. Blood stream infection in ICU (post randomisation) defined using the Center for Disease Control and Prevention/National Healthcare Safety Network criteria
6. Length of stay in ICU and in hospital post randomisation
7. Febrile non-haemolytic transfusion reactions
8. EQ-5D score at Day 90 post randomisation

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalised in ICU with an anticipated ICU stay of at least 24 hours, in whom the decision has been made by medical staff to transfuse at least one RBC unit.

Exclusion Criteria:

* Age younger than 18
* Previous RBC transfusion during the current hospital admission (including transfusion in another hospital for transferred patients)
* Diagnosis of transplantation or hematologic diseases
* Pregnancy
* Cardiac surgery during the present hospital admission
* Expected to die imminently (<24hrs)
* The treating physician believes it is not in the best interest of the patient to be randomised in this trial.
* Known objection to the administration of human blood products
* Participation in a competing study (see below)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4994 (Actual)
Dates: Start 2012-10; Primary Completion 2017-04 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D. James Cooper, A.O., M.D., Principal Investigator — Monash University/Alfred Hospital
Locations (60):
- Australia (42):
  - The Alfred Hospital, Melbourne, Victoria
  - Lyell McEwin Hospital, Adelaide
  - Queen Elizabeth Hospital, Adelaide
  - Royal Adelaide Hospital, Adelaide
  - Albury Hospital, Albury
  - Bendigo Hospital, Bendigo
  - Logan Hospital, Brisbane
  - Mater Adult Hospital, Brisbane
  - Mater Private Hospital, Brisbane
  - Princess Alexandra Hospital, Brisbane
  - Royal Brisbane and Women's Hospital, Brisbane
  - Calvary Health, Canberra
  - Canberra Hospital, Canberra
  - Dandenong Hospital, Dandenong
  - Geelong Hospital, Geelong
  - Gold Coast Hospital, Gold Coast
  - Gosford Hospital, Gosford
  - Austin Hospital, Heidelberg
  - Royal Hobart Hospital, Hobart
  - Cabrini Hospital, Melbourne
  - Frankston Hospital, Melbourne
  - Knox Private Hospital, Melbourne
  - Monash Medical Centre, Melbourne
  - Northern Hospital, Melbourne
  - Royal Melbourne Hospital, Melbourne
  - St Vincent's Hospital, Melbourne
  - Sunshine Hospital, Melbourne
  - Western Hospital, Melbourne
  - Calvary Mater Newcastle, Newcastle
  - John Hunter Hospital, Newcastle
  - Fiona Stanley Hospital, Perth
  - Royal Perth Hospital, Perth
  - St John of God Murdoch Hospital, Perth
  - Epworth Hospital, Richmond
  - Blacktown Hospital, Sydney
  - Nepean Hospital, Sydney
  - Prince of Wales Hospital, Sydney
  - Royal Prince Alfred Hospital, Sydney
  - St George Hospital, Sydney
  - St Vincent's Hospital, Sydney
  - Tamworth Hospital, Tamworth
  - Wollongong Hospital, Wollongong
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Tampere University Hospital, Tampere
- Ireland (6):
  - Cork University Hospital, Cork
  - Beaumont Hospital, Dublin
  - St James's Hospital, Dublin
  - St Vincent's University Hospital, Dublin
  - Galway Regional Hospital, Galway
  - Limerick Regional Hospital, Limerick
- New Zealand (9):
  - Auckland City Hospital CVICU, Auckland
  - Auckland City Hospital DCCM, Auckland
  - Middlemore Hospital, Auckland
  - North Shore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Nelson Hospital, Nelson
  - Wellington Hospital, Wellington
- King Abdulaziz Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Radford M, Estcourt LJ, Sirotich E, Pitre T, Britto J, Watson M, Brunskill SJ, Fergusson DA, Doree C, Arnold DM. Restrictive versus liberal red blood cell transfusion strategies for people with haematological malignancies treated with intensive chemotherapy or radiotherapy, or both, with or without haematopoietic stem cell support. Cochrane Database Syst Rev. 2024 May 23;5(5):CD011305. doi: 10.1002/14651858.CD011305.pub3. PMID 38780066
- [Derived] Cooper DJ, McQuilten ZK, Nichol A, Ady B, Aubron C, Bailey M, Bellomo R, Gantner D, Irving DO, Kaukonen KM, McArthur C, Murray L, Pettila V, French C; TRANSFUSE Investigators and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Age of Red Cells for Transfusion and Outcomes in Critically Ill Adults. N Engl J Med. 2017 Nov 9;377(19):1858-1867. doi: 10.1056/NEJMoa1707572. Epub 2017 Sep 27. PMID 28952891
- [Derived] Kaukonen KM, Bailey M, Ady B, Aubron C, French C, Gantner D, Irving D, Murray L, Nichol A, Pettila V, McQuilten Z, Cooper DJ. A randomised controlled trial of standard transfusion versus fresher red blood cell use in intensive care (TRANSFUSE): protocol and statistical analysis plan. Crit Care Resusc. 2014 Dec;16(4):255-61. PMID 25437218
- [Derived] Kekre N, Mallick R, Allan D, Tinmouth A, Tay J. The impact of prolonged storage of red blood cells on cancer survival. PLoS One. 2013 Jul 16;8(7):e68820. doi: 10.1371/journal.pone.0068820. Print 2013. PMID 23874777

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm B (Short Term Storage): Blood Transfusion Freshest blood.
  Blood transfusion: Blood transfusion in ICU patients aged 18 and over.
- Standard of Care (Long-term Storage): Blood Transfusion Standard of care- oldest blood.
  Blood transfusion: Blood transfusion in ICU patients aged 18 and over.
Period: Overall Study
Arm/Group | Arm B (Short Term Storage) | Standard of Care (Long-term Storage)
Started | 2490 | 2504
Completed | 2457 | 2462
Not Completed | 33 | 42

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care (Long Term Storage): Blood Transfusion Standard of care- oldest blood.
  Blood transfusion: Blood transfusion in ICU patients aged 18 and over.
- Total: Total of all reporting groups
Arm/Group | Arm B (Short Term Storage) | Standard of Care (Long Term Storage) | Total
Number analyzed (Participants) | 2457 | 2462 | 4919
Age, Continuous [Median (Standard Deviation); unit: years] | 62.5 (16.8) | 61.4 (17.3) | 62.0 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1146 | 1204 | 2350
  Male | 1311 | 1258 | 2569
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Primary Diagnosis [Count of Participants; unit: Participants]
  Cardiovascular Condition | 326 | 342 | 668
  Gastrointestinal Condition | 551 | 514 | 1065
  Respiratory Condition | 413 | 422 | 835
  Sepsis | 413 | 396 | 809
  Trauma | 240 | 262 | 502
  Neurological Condition | 177 | 195 | 372
  Metabolic Condition | 68 | 71 | 139
  Musculoskeletal | 103 | 110 | 213
  Renal Condition | 110 | 109 | 219
  Other Condition | 51 | 35 | 86
  Missing Condition | 5 | 6 | 11
APACHE III [Median (Standard Deviation); unit: units on a scale] — The APACHE III score consists of several parts including the primary reason for ICU admission, age, sex, race, pre existing comorbidities, and location prior to ICU admission. The range of APACHE III score is from 0 to 299 points. APACHE III is widely used to assess illness severity of patients admitted to ICU and to compare risk-adjusted outcomes between ICUs. Increasing score is associated with increasing risk of hospital death. A score of 0 is associated with a very low risk of death
  units on a scale | 72.6 (29.2) | 73.2 (29.6) | 72.9 (29.4)
ABO Blood group [Count of Participants; unit: Participants]
  Group A | 928 | 961 | 1889
  Group B | 310 | 303 | 613
  Group O | 1126 | 1105 | 2231
  Group AB | 92 | 93 | 185
  Missing Data | 1 | 0 | 1
Haemoglobin at Admission to ICU [Median (Standard Deviation); unit: g/liter] | 102 (23.1) | 102 (23.6) | 102 (23.3)
Haemoglobin at randomisation [Median (Standard Deviation); unit: g/liter] | 77.4 (12.8) | 77.3 (13.0) | 77.3 (12.9)
SOFA Score [Median (Inter-Quartile Range); unit: units on a scale] — The Sequential Organ Failure Assessment (SOFA) Score is a mortality prediction score that is based on the degree of dysfunction of six organ systems. The score was calculated on admission.
  The SOFA scoring system is useful in predicting the clinical outcomes of critically ill patient.
  The SOFA score ranges from 0-24. A score of 0 predicts a very good outcome. A score of 24 predicts a very poor patient outcome
  units on a scale | 7 [4 to 10] | 7 [5 to 10] | 7 [5 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Mortality at Day 90
Description: Mortality at Day 90
Time Frame: 90 Day
Population: Pre specified Sub groups
Measure: Number; unit: participants
Arm/Group | Arm B (Short Term Storage) | Standard of Care (Long Term Storage)
Number analyzed (Participants) | 2457 | 2462
participants
  All patients | 610 | 594
  Group O: number analyzed (Participants) | 1126 | 1105
  Group O | 264 | 259
  Non-Group O: number analyzed (Participants) | 1330 | 1357
  Non-Group O | 346 | 335
  APACHE III risk of Death <21.5%: number analyzed (Participants) | 1243 | 1209
  APACHE III risk of Death <21.5% | 152 | 169
  APACHE III risk of Death =or>21.5%: number analyzed (Participants) | 1212 | 1251
  APACHE III risk of Death =or>21.5% | 457 | 425
  Baseline SOFA score = or < 7: number analyzed (Participants) | 1317 | 1273
  Baseline SOFA score = or < 7 | 210 | 191
  Baseline SOFA score >7: number analyzed (Participants) | 1140 | 1189
  Baseline SOFA score >7 | 400 | 403

2. Secondary Outcome: Mortality at Day 28
Description: Mortality at day 28
Time Frame: 28 day
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B (Short Term Storage) | Standard of Care (Long Term Storage)
Number analyzed (Participants) | 2457 | 2462
Participants | 476 | 463

3. Secondary Outcome: Persistent Organ Dysfunction Combined With Death Measured at Day 28
Description: Persistent Organ Dysfunction combined with death measured at day 28
Time Frame: day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B (Short Term Storage) | Standard of Care (Long Term Storage)
Number analyzed (Participants) | 2457 | 2462
Participants | 573 | 549

4. Secondary Outcome: Days Alive and Free of Mechanical Ventilation
Description: Days alive and free of mechanical ventilation
Time Frame: day 28
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Arm B (Short Term Storage) | Standard of Care (Long Term Storage)
Number analyzed (Participants) | 2457 | 2462
days | 25 [11 to 28] | 25 [13 to 28]

5. Secondary Outcome: Day Alive and Free of Renal Replacement Therapy.
Description: Day alive and free of renal replacement therapy.
Time Frame: day 28
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Arm B (Short Term Storage) | Standard of Care (Long Term Storage)
Number analyzed (Participants) | 2457 | 2462
days | 28 [22 to 28] | 22 [22 to 28]

6. Secondary Outcome: Blood Stream Infection in ICU (Post Randomisation)
Description: Blood stream infection in ICU (post randomisation) Time Frame is in Days
Time Frame: While in ICU-Median duration in ICU - short term storage group was 4.2 days (2.0 - 9.3), long term storage group was 4.2 days (1.9 - 9.4)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B (Short Term Storage) | Standard of Care (Long-term Storage)
Number analyzed (Participants) | 2457 | 2462
Participants | 123 | 88

7. Secondary Outcome: Length of Stay in ICU and in Hospital Post Randomisation (Days)
Description: Median duration in ICU - short term storage group was 4.2 (2.0 - 9.3), long term storage group was 4.2 (1.9 - 9.4) Median duration in Hospital - short term storage group was 14.5 (7.4 - 27.5), long term storage group was 14.7 (7.4 - 28.3) In Days
Time Frame: Median duration in ICU- short term storage group 4.2 Days (2.0 - 9.3), long term storage group 4.2 Days (1.9 - 9.4). Median duration in Hospital- short term storage group was 14.5 days (7.4 - 27.5), long term storage group was 14.7 days(7.4 - 28.3)
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Arm B (Short Term Storage) | Standard of Care (Long Term Storage)
Number analyzed (Participants) | 2457 | 2462
Days
  Days in ICU | 4.2 [2.0 to 9.3] | 4.2 [1.9 to 9.4]
  Days in Hospital | 14.5 [7.4 to 27.5] | 14.7 [7.4 to 28.3]

8. Secondary Outcome: Proportion of Patients Who Suffer at Least One Febrile Non-haemolytic Transfusion Reaction in ICU
Description: Proportion of patients who suffer at least one febrile non-haemolytic transfusion reaction in ICU
Time Frame: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Arm B (Short Term Storage) | Standard of Care (Long-term Storage)
Number analyzed (Participants) | 2457 | 2462
Participants | 35 | 39

9. Secondary Outcome: EuroQol-5Dimension 5 Level (EQ-5D-5L) Score at Day 180 Post Randomisation
Description: EuroQol-5Dimension 5 level (EQ-5D-5L) score at day 180 post randomisation - not reported yet
Time Frame: Day 180
Reporting Status: Not Posted, anticipated posting 2022-07

ADVERSE EVENTS:
Time Frame: Primary outcome was all-cause mortality measured up to day 90. Secondary outcomes included mortality / persistent organ dysfunction or death / days alive and free of mechanical ventilation / days alive and free of renal-replacement therapy measured all measured at day 28, new bloodstream infection measured during ICU stay, febrile nonhemolytic transfusion reactions during ICU stay, length of stay (hospital and ICU), and quality of life measured at day 180 after randomization.
Description: We defined a febrile nonhemolytic transfusion reaction as occurring when a patient had an unexpected increase in temperature of 1°C or more within 4 hours after transfusion in the absence of other pyretic stimuli.
Arm/Group | Arm B (Short Term Storage) | Standard of Care (Long Term Storage)
All-Cause Mortality (participants affected / at risk) | 687/2410 | 678/2414
Serious Adverse Events (participants affected / at risk) | 0/2457 | 0/2462
Other Adverse Events (participants affected / at risk) | 158/2457 | 127/2462
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm B (Short Term Storage) (N=2457) | Standard of Care (Long Term Storage) (N=2462)
Febrile Nonhaemolytic transfusion reaction (Immune system disorders) | 35 | 39
New Bloodstream Infection in ICU (Blood and lymphatic system disorders) | 123 | 88

LIMITATIONS AND CAVEATS:
The red-cell age in each treatment group was not prespecified but was determined by the blood-bank inventory at each institution.

We did not design the trial to assign red cells toward the end of their shelf life (35 to 42 days).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-11-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT01638416/Prot_SAP_000.pdf
  • Informed Consent Form (2013-06-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT01638416/ICF_001.pdf